CLINICAL TRIAL: NCT01149421
Title: The Effect of LY2189265 on Blood Pressure and Heart Rate, as Assessed by Ambulatory Blood Pressure Monitoring, in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of the Effect of LY2189265 on Blood Pressure and Heart Rate in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13631; H9X-MC-GBDN (Other: Eli Lilly and Company); CTRI/2010/091/001444 (Registry Identifier: Clinical Trials Register India)
Record Dates: First submitted 2010-06-15; First posted 2010-06-23 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Diabetes; Ambulatory Blood Pressure Monitoring; ABPM; Blood Pressure; Heart Rate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.5 milligram (mg) LY2189265 (Experimental): LY2189265: 1.5 milligram (mg), subcutaneous (SC), once weekly (QW)
  Interventions: Drug: LY2189265
- 0.75 milligram (mg) LY2189265 (Experimental): LY2189265: 0.75 milligram (mg), subcutaneous (SC), once weekly (QW)
  Interventions: Drug: LY2189265
- Placebo (Placebo Comparator): Placebo: subcutaneous (SC), once weekly (QW)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2189265 — Administered as a subcutaneous injection once weekly for 26 weeks
  Other Names: Dulaglutide
  Arms: 0.75 milligram (mg) LY2189265; 1.5 milligram (mg) LY2189265
Drug: Placebo — Administered as a subcutaneous injection once weekly for 26 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of 2 doses of LY2189265 on blood pressure and heart rate using 24-hour ambulatory blood pressure monitoring (ABPM), in participants with type 2 diabetes mellitus treated with oral antihyperglycemic medications (OAMs).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes taking 1 or more oral diabetes medications and have taken these medications for at least 1 month prior to screening
* Glycosylated hemoglobin (HbA1c) value ≥7% and ≤9.5% at screening
* Mean blood pressure >90/60 millimeters of mercury (mmHg) and <140/90 mmHg at screening
* If treated for hypertension, are taking 3 or less antihypertensive medications and have been taking these medications for at least 1 month prior to screening
* Stable weight for 3 months prior to screening
* Body mass index (BMI) greater than or equal to 23 kilogram-meter squared (kg/m^2)
* Willing to wear an ambulatory blood pressure monitoring device for at least 24 hours on multiple occasions
* Women of childbearing potential must test negative for pregnancy and be willing to use a reliable method of birth control
* Male participants must use a reliable method of birth control

Exclusion Criteria:

* Myocardial infarction, stroke, or hospitalization for heart failure within 3 months prior to screening, or heart failure Class III or IV at screening
* Ongoing or history of frequent intermittent tachyarrhythmia
* Resting heart rate <60 beats per minute (bpm) or >100 bpm at screening
* Work rotating shifts or work during the hours of 2200 to 0700
* Chronic insulin therapy
* Use of a glucagon-like peptide 1 (GLP-1) receptor agonist within 3 months prior to screening, or a dipeptidylpeptidase-IV (DPP-IV) inhibitor within 2 weeks prior to screening
* Nondominant arm circumference >42 centimeter (cm)
* Use of drugs to promote weight loss
* Chronic use of systemic steroids
* Gastric emptying abnormality or bariatric surgery
* Hepatitis, other liver disease, or alanine transaminase (ALT) >3 times the upper limit of normal
* Acute or chronic pancreatitis
* Severe renal impairment
* Active autoimmune disease or uncontrolled endocrine abnormality
* Self or family history of thyroid cancer, medullary C-cell hyperplasia, or type 2A or 2B multiple endocrine neoplasia
* Calcitonin value greater than or equal to 20 picograms per milliliter (pg/ml) at screening
* Transplanted organ except corneal transplants
* Active or untreated cancer or in remission <5 years, except skin, in situ cervical, or prostate cancer
* Sickle-cell disease, hemolytic anemia, or another hematological condition that may interfere with HbA1c testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (76):
- United States (42):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Gables, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Haven, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cartersville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucker, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paducah, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auburn, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jefferson City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jefferson Hills, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Georgetown, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
- Argentina (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Fe
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Red Deer, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. John's, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakville, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laval, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Laurent, Quebec
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., České Budějovice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Český Krumlov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Přerov
- Denmark (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ballerup Municipality
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vejle
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbatore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludhiana
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce

REFERENCES:
- [Derived] Ferdinand KC, Dunn J, Nicolay C, Sam F, Blue EK, Wang H. Weight-dependent and weight-independent effects of dulaglutide on blood pressure in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):49. doi: 10.1186/s12933-023-01775-x. PMID 36894938

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.5 Milligram (mg) LY2189265: LY2189265: 1.5 milligram (mg), subcutaneous (SC), once weekly (QW) for 26 weeks
- 0.75 Milligram (mg) LY2189265: LY2189265: 0.75 milligram (mg), subcutaneous (SC), once weekly (QW) for 26 weeks
- Placebo: Placebo: subcutaneous (SC), once weekly (QW) for 26 weeks
Period: Overall Study
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Started | 251 | 254 | 250
Received at Least One Dose of Study Drug | 251 | 254 | 250
Completed | 199 | 225 | 206
Not Completed | 52 | 29 | 44
Not completed — Adverse Event | 22 | 6 | 11
Not completed — Withdrawal by Subject | 20 | 12 | 13
Not completed — Sponsor Decision | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 4 | 5
Not completed — Physician Decision | 5 | 3 | 6
Not completed — Entry Criteria Not Met | 1 | 1 | 2
Not completed — Protocol Violation | 2 | 2 | 6

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of LY2189265 or Placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo | Total
Number analyzed (Participants) | 251 | 254 | 250 | 755
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.96 (10.14) | 57.05 (10.17) | 56.43 (10.50) | 56.48 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 123 | 119 | 363
  Male | 130 | 131 | 131 | 392
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 101 | 91 | 287
  Not Hispanic or Latino | 156 | 153 | 159 | 468
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 22 | 24 | 23 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 23 | 21 | 22 | 66
  White | 201 | 204 | 203 | 608
  More than one race | 3 | 5 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 132 | 137 | 139 | 408
  Czech Republic | 12 | 12 | 13 | 37
  Puerto Rico | 12 | 14 | 14 | 40
  Canada | 34 | 32 | 30 | 96
  Argentina | 29 | 28 | 25 | 82
  Brazil | 8 | 6 | 7 | 21
  Denmark | 9 | 11 | 8 | 28
  India | 15 | 14 | 14 | 43
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 32.80 (5.66) | 32.55 (5.86) | 33.53 (6.49) | 32.96 (6.02)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7.93 (0.76) | 7.91 (0.73) | 7.94 (0.78) | 7.93 (0.76)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 90.42 (18.58) | 90.45 (18.74) | 93.90 (21.26) | 91.58 (19.60)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 7.61 (5.30) | 8.99 (6.39) | 8.40 (5.76) | 8.34 (5.86)
Mean Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Clinic systolic blood pressure (SBP) measurements were taken in triplicate after the participant was seated for 5 minutes using an automated digital professional blood pressure monitor. The mean of the last 2 clinic readings at screening determined study eligibility; the mean of 3 readings at baseline and all post-baseline visits was used for analyses.
  millimeters of mercury (mmHg)
    Mean 24-hour Systolic Blood Pressure | 130.85 (12.14) | 132.08 (12.97) | 131.13 (11.23) | 131.36 (12.13)
    Mean Daytime Systolic Blood Pressure | 133.92 (12.30) | 135.37 (13.36) | 134.15 (11.70) | 134.48 (12.48)
    Mean Nighttime Systolic Blood Pressure | 121.68 (14.39) | 122.10 (14.83) | 121.92 (12.82) | 121.90 (14.02)
    Mean Seated Systolic Blood Pressure (Clinic) | 126.71 (12.44) | 127.42 (12.79) | 126.81 (13.67) | 126.98 (12.96)
Mean Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Clinic diastolic blood pressure (DBP) measurements were taken in triplicate after the participant was seated for 5 minutes using an automated digital professional blood pressure monitor. The mean of the last 2 clinic readings at screening determined study eligibility; the mean of 3 readings at baseline and all post-baseline visits was used for analyses.
  millimeters of mercury (mmHg)
    Mean 24-hour Diastolic Blood Pressure | 76.29 (8.39) | 76.64 (8.38) | 75.96 (7.79) | 76.30 (8.18)
    Mean Daytime Diastolic Blood Pressure | 78.93 (8.77) | 79.35 (8.81) | 78.68 (8.27) | 78.99 (8.61)
    Mean Nighttime Diastolic Blood Pressure | 68.83 (9.70) | 68.92 (9.47) | 68.21 (8.70) | 68.65 (9.29)
    Mean Seated Diastolic Blood Pressure (Clinic) | 75.95 (8.61) | 75.81 (8.84) | 76.14 (9.19) | 75.97 (8.87)
Mean Heart Rate (HR) [Mean (Standard Deviation); unit: beats per minute (bpm)] — Clinic heart rate (HR) measurements were taken in triplicate after the participant was seated for 5 minutes using an automated digital professional blood pressure monitor. The mean of the last 2 clinic readings at screening determined study eligibility; the mean of 3 readings at baseline and all post-baseline visits was used for analyses.
  beats per minute (bpm)
    Mean 24-Hour Heart Rate | 79.86 (10.83) | 79.01 (9.75) | 79.91 (9.97) | 79.59 (10.18)
    Mean Daytime Heart Rate | 82.47 (11.61) | 81.99 (10.45) | 82.96 (10.69) | 82.47 (10.92)
    Mean Nighttime Heart Rate | 72.78 (10.76) | 71.33 (9.94) | 72.20 (10.35) | 72.10 (10.36)
    Mean Seated Heart Rate (Clinic) | 74.50 (10.81) | 73.71 (9.31) | 74.90 (10.56) | 74.37 (10.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 16 Weeks in Mean 24-hour Systolic Blood Pressure (SBP)
Description: Mean 24-hour systolic blood pressure (SBP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg) | -3.41 (0.61) | -1.70 (0.58) | -0.63 (0.59)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — P-value reported for non-inferior to Placebo. The adjustment for multiplicity was based on a tree-gatekeeping testing strategy; Least Squares Mean Difference = -2.79, 97.3% CI 2-sided [-4.58 to -1.00]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.07, 97.3% CI 2-sided [-2.83 to 0.68]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Since non-inferiority was confirmed, superiority analysis was pursued. P-value reported for superior to Placebo. The adjustment for multiplicity was based on a tree-gatekeeping testing strategy
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.149, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 3]

2. Secondary Outcome: Change From Baseline to 26 Weeks in Mean 24-hour Systolic Blood Pressure (SBP)
Description: as for outcome 1
Time Frame: Baseline, 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable systolic blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg) | -2.51 (0.63) | -1.56 (0.60) | 0.15 (0.62)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.66, 97.3% CI 2-sided [-4.53 to -0.79]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.71, 97.3% CI 2-sided [-3.54 to 0.12]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.36, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 3]

3. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean 24-hour Diastolic Blood Pressure (DBP)
Description: Mean 24-hour diastolic blood pressure (DBP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means of change from baseline was analyzed using mixed model repeated measures (MMRM) adjusted by baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable diastolic blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)]
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg)]
  Mean 24-Hour, Week 16 | -0.23 (0.38) | -0.13 (0.37) | -0.55 (0.37)
  Mean 24-Hour, Week 26 | 0.26 (0.40) | -0.09 (0.38) | -0.24 (0.39)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — Treatment comparison at 16 weeks. P-value reported for non-inferior to Placebo. The adjustment for multiplicity was based on a tree-gatekeeping testing strategy; Least Squares Mean Difference = 0.32, 97.3% CI 2-sided [-0.80 to 1.43]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean Difference = 0.42, 97.3% CI 2-sided [-0.67 to 1.52]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.870, Mixed Models Analysis — Treatment comparison at 16 weeks. Since non-inferiority was confirmed, superiority analysis was pursued. P-value reported for superior to Placebo. The adjustment for multiplicity was based on a tree-gatekeeping testing strategy
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.915, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks. P-value reported for non-inferior to Placebo. The adjustment for multiplicity was based on a tree-gatekeeping testing strategy; Least Squares Mean Difference = 0.50, 97.3% CI 2-sided [-0.68 to 1.68]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 5]; Least Squares Mean Difference = 0.16, 97.3% CI 2-sided [-1.00 to 1.31]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.929, Mixed Models Analysis — Treatment comparison at 26 weeks. Since non-inferiority was confirmed, superiority analysis was pursued. P-value reported for superior to Placebo. The adjustment for multiplicity was based on a tree-gatekeeping testing strategy
Statistical Analysis 8: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.776, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 7]

4. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean 24-Hour Heart Rate (HR)
Description: Mean 24-hour heart rate (HR) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Heart rate measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable heart rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
beats per minute (bpm)
  Mean 24-Hour HR, Week 16 | 3.70 (0.45) | 2.48 (0.43) | 0.86 (0.44)
  Mean 24-Hour HR, Week 26 | 4.18 (0.47) | 1.94 (0.46) | 0.68 (0.47)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p = 0.556, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean Difference = 2.84, 97.3% CI 2-sided [1.52 to 4.16]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p = 0.018, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least Squares Mean Difference = 1.62, 97.3% CI 2-sided [0.32 to 2.92]
Statistical Analysis 3: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 1.00, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p = 0.904, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 5]; Least Squares Mean Difference = 3.50, 97.3% CI 2-sided [2.10 to 4.91]
Statistical Analysis 5: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Non-Inferiority or Equivalence — If non-inferiority was confirmed, then superiority analysis was pursued; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 5]; Least Squares Mean Difference = 1.26, 97.3% CI 2-sided [-0.13 to 2.64]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.996, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 7]

5. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean 24-hour Pulse Pressure
Description: Mean 24-hour pulse pressure (PP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Pulse pressure (PP) measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable pulse pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg)
  Mean 24-Hour PP, Week 16 | -3.07 (0.36) | -1.60 (0.35) | -0.02 (0.36)
  Mean 24-Hour PP, Week 26 | -2.64 (0.38) | -1.53 (0.37) | 0.46 (0.37)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 16 weeks; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-4.00 to -2.09]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — Treatment comparison at 16 weeks; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-2.51 to -0.64]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks; Mean Difference (Final Values) = -3.10, 95% CI 2-sided [-4.10 to -2.09]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-2.98 to -1.00]

6. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean 24-hour Mean Arterial Pressure (MAP)
Description: Mean 24-hour mean arterial pressure (MAP) was measured by a using 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable mean arterial pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg)
  Week 16 | -1.31 (0.43) | -0.65 (0.42) | -0.60 (0.42)
  Week 26 | -0.74 (0.44) | -0.57 (0.42) | -0.15 (0.43)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.218, Mixed Models Analysis — Treatment comparison at 16 weeks; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.84 to 0.42]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.931, Mixed Models Analysis — Treatment comparison at 16 weeks; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-1.16 to 1.06]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.315, Mixed Models Analysis — Treatment comparison at 26 weeks; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.72 to 0.55]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.465, Mixed Models Analysis — Treatment comparison at 26 weeks; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.54 to 0.70]

7. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean Daytime, Nighttime, and Clinic Systolic Blood Pressure (SBP)
Description: Mean daytime and nighttime systolic blood pressure (SBP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension. Clinic SBP was measured in the clinic using the Omron HEM 907XL Blood Pressure monitor.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable systolic blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
millimeters of mercury (mmHg)
  Mean Daytime SBP, Week 16 (n=247, n=251, n=249) | -3.67 (0.66) | -1.57 (0.63) | -0.34 (0.64)
  Mean Daytime SBP, Week 26 (n=247, n=251, n=249) | -2.52 (0.68) | -1.47 (0.65) | 0.35 (0.67)
  Mean Nighttime SBP, Week 16 (n=247, n=251, n=249) | -2.32 (0.76) | -1.23 (0.73) | -1.08 (0.74)
  Mean Nighttime SBP, Week 26 (n=247, n=251, n=249) | -2.40 (0.75) | -1.43 (0.72) | -0.05 (0.73)
  Mean Clinic SBP, Week 16 (n=251, n=254, n=250) | -2.33 (0.75) | -1.26 (0.72) | -0.73 (0.73)
  Mean Clinic SBP, Week 26 (n=251, n=254, n=250) | -2.29 (0.77) | -0.74 (0.74) | 0.40 (0.75)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime systolic blood pressure (SBP) at 16 weeks; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-5.04 to -1.61]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.153, Mixed Models Analysis — Treatment comparison of mean daytime systolic blood pressure (SBP) at 16 weeks; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-2.91 to 0.46]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Treatment comparison of mean daytime systolic blood pressure (SBP) at 26 weeks; Mean Difference (Final Values) = -2.87, 95% CI 2-sided [-4.66 to -1.09]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis — Treatment comparison of mean daytime systolic blood pressure (SBP) at 26 weeks; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-3.57 to -0.07]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.221, Mixed Models Analysis — Treatment comparison of mean nighttime systolic blood pressure (SBP) at 16 weeks; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-3.23 to 0.75]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.884, Mixed Models Analysis — Treatment comparison of mean nighttime systolic blood pressure (SBP) at 16 weeks; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-2.10 to 1.81]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis — Treatment comparison of mean nighttime systolic blood pressure (SBP) at 26 weeks; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-4.31 to -0.39]
Statistical Analysis 8: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.159, Mixed Models Analysis — Treatment comparison of mean nighttime systolic blood pressure (SBP) at 26 weeks; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-3.31 to 0.54]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.122, Mixed Models Analysis — Treatment comparison of mean clinic systolic blood pressure (SBP) at 16 weeks
Statistical Analysis 10: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.601, Mixed Models Analysis — Treatment comparison of mean clinic systolic blood pressure (SBP) at 16 weeks
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — Treatment comparison of mean clinic systolic blood pressure (SBP) at 26 weeks
Statistical Analysis 12: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.274, Mixed Models Analysis — Treatment comparison of mean clinic systolic blood pressure (SBP) at 26 weeks

8. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean Daytime, Nighttime, and Clinic Diastolic Blood Pressure (DBP)
Description: Mean daytime and nighttime diastolic blood pressure (DBP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means of change from baseline was analyzed using mixed model repeated measures (MMRM) adjusted by baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension. Clinic DBP was measured in the clinic using the Omron HEM 907XL Blood Pressure monitor.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable diastolic blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
millimeters of mercury (mmHg)
  Mean Daytime DBP, Week 16 (n=247, n=251, n=249) | -0.09 (0.43) | 0.14 (0.41) | -0.30 (0.42)
  Mean Daytime DBP, Week 26 (n=247, n=251, n=249) | 0.52 (0.43) | 0.08 (0.41) | -0.07 (0.42)
  Mean Nighttime DBP, Week 16 (n=247, n=251, n=249) | -0.01 (0.49) | -0.28 (0.48) | -1.10 (0.48)
  Mean Nighttime DBP, Week 26 (n=247, n=251, n=249) | -0.22 (0.51) | -0.42 (0.50) | -0.69 (0.51)
  Mean Clinic DBP, Week 16 (n=251, n=254, n=250) | -0.21 (0.52) | 0.76 (0.50) | -0.21 (0.51)
  Mean Clinic DBP, Week 26 (n=251, n=254, n=250) | 0.59 (0.50) | 0.69 (0.48) | 0.61 (0.49)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.717, Mixed Models Analysis — Treatment comparison of mean daytime diastolic blood pressure (DBP) at 16 weeks; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.91 to 1.32]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.427, Mixed Models Analysis — Treatment comparison of mean daytime diastolic blood pressure (DBP) at 16 weeks; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.65 to 1.54]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.300, Mixed Models Analysis — Treatment comparison of mean daytime diastolic blood pressure (DBP) at 26 weeks; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-0.53 to 1.73]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.788, Mixed Models Analysis — Treatment comparison of mean daytime diastolic blood pressure (DBP) at 26 weeks; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.96 to 1.26]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.098, Mixed Models Analysis — Treatment comparison of mean nighttime diastolic blood pressure (DBP) at 16 weeks; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [-0.20 to 2.37]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.203, Mixed Models Analysis — Treatment comparison of mean nighttime diastolic blood pressure (DBP) at 16 weeks; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.44 to 2.08]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.493, Mixed Models Analysis — Treatment comparison of mean nighttime diastolic blood pressure (DBP) at 26 weeks; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.88 to 1.82]
Statistical Analysis 8: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis — Treatment comparison of mean nighttime diastolic blood pressure (DBP) at 26 weeks; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-1.06 to 1.60]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.990, Mixed Models Analysis — Treatment comparison of mean clinic diastolic blood pressure (DBP) at 16 weeks
Statistical Analysis 10: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.173, Mixed Models Analysis — Treatment comparison of mean clinic diastolic blood pressure (DBP) at 16 weeks
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.972, Mixed Models Analysis — Treatment comparison of mean clinic diastolic blood pressure (DBP) at 26 weeks
Statistical Analysis 12: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.904, Mixed Models Analysis — Treatment comparison of mean clinic diastolic blood pressure (DBP) at 26 weeks

9. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean Daytime, Nighttime, and Clinic Heart Rate (HR)
Description: Daytime and nighttime heart rate (HR) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Heart rate measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension. Clinic HR was measured in the clinic using the Omron HEM 907XL Blood Pressure monitor.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable heart rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
beats per minute (bpm)
  Mean Daytime HR, Week 16 (n=247, n=251, n=249) | 3.56 (0.50) | 2.22 (0.49) | 1.07 (0.49)
  Mean Daytime HR, Week 26 (n=247, n=251, n=249) | 4.24 (0.51) | 1.59 (0.49) | 0.67 (0.50)
  Mean Nighttime HR, Week 16 (n=247, n=251, n=249) | 4.60 (0.51) | 3.43 (0.49) | 0.65 (0.50)
  Mean Nighttime HR, Week 26 (n=247, n=251, n=249) | 4.76 (0.57) | 3.01 (0.54) | 0.77 (0.55)
  Mean Clinic HR, Week 16 (n=251, n=254, n=250) | 3.97 (0.49) | 2.11 (0.48) | 0.46 (0.48)
  Mean Clinic HR, Week 26 (n=251, n=254, n=250) | 4.89 (0.54) | 1.93 (0.52) | -0.11 (0.53)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime heart rate (HR) at 16 weeks; Mean Difference (Final Values) = 2.49, 95% CI 2-sided [1.17 to 3.80]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis — Treatment comparison of mean daytime heart rate (HR) at 16 weeks; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-0.14 to 2.45]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime heart rate (HR) at 26 weeks; Mean Difference (Final Values) = 3.57, 95% CI 2-sided [2.23 to 4.91]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.168, Mixed Models Analysis — Treatment comparison of mean daytime heart rate (HR) at 26 weeks; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-0.39 to 2.24]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean nighttime heart rate (HR) at 16 weeks; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [2.62 to 5.28]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean nighttime heart rate (HR) at 16 weeks; Mean Difference (Final Values) = 2.78, 95% CI 2-sided [1.47 to 4.09]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean nighttime heart rate (HR) at 26 weeks; Mean Difference (Final Values) = 3.98, 95% CI 2-sided [2.49 to 5.47]
Statistical Analysis 8: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Treatment comparison of mean nighttime heart rate (HR) at 26 weeks; Mean Difference (Final Values) = 2.24, 95% CI 2-sided [0.78 to 3.70]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean clinic heart rate (HR) at 16 weeks
Statistical Analysis 10: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — Treatment comparison of mean clinic heart rate (HR) at 16 weeks
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean clinic heart rate (HR) at 26 weeks
Statistical Analysis 12: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — Treatment comparison of mean clinic heart rate (HR) at 26 weeks

10. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean Daytime and Nighttime Pulse Pressure
Description: Mean daytime and nighttime pulse pressure (PP) was measured by using a 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Pulse pressure (PP) measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable pulse pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg)
  Mean Daytime PP, Week 16 | -3.46 (0.40) | -1.76 (0.38) | 0.01 (0.39)
  Mean Daytime PP, Week 26 | -2.90 (0.42) | -1.62 (0.41) | 0.51 (0.42)
  Mean Nighttime PP, Week 16 | -2.23 (0.45) | -0.92 (0.43) | 0.02 (0.44)
  Mean Nighttime PP, Week 26 | -2.09 (0.43) | -0.96 (0.41) | 0.65 (0.42)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime pulse pressure (PP) at 16 weeks; Mean Difference (Final Values) = -3.47, 95% CI 2-sided [-4.50 to -2.43]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime pulse pressure (PP) at 16 weeks; Mean Difference (Final Values) = -1.77, 95% CI 2-sided [-2.79 to -0.75]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime pulse pressure (PP) at 26 weeks; Mean Difference (Final Values) = -3.40, 95% CI 2-sided [-4.52 to -2.28]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean daytime pulse pressure (PP) at 26 weeks; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-3.23 to -1.03]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean nighttime pulse pressure (PP) at 16 weeks; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-3.43 to -1.07]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.113, Mixed Models Analysis — Treatment comparison of mean nighttime pulse pressure (PP) at 16 weeks; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.09 to 0.22]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of mean nighttime pulse pressure (PP) at 26 weeks; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-3.86 to -1.62]
Statistical Analysis 8: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — Treatment comparison of mean nighttime pulse pressure (PP) at 26 weeks; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-2.72 to -0.51]

11. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Mean Daytime and Nighttime Mean Arterial Pressure (MAP)
Description: Mean daytime and nighttime mean arterial pressure (MAP) was measured by a using 24-hour ambulatory blood pressure monitoring (ABPM) device attached to the participant's nondominant arm. Ambulatory blood pressure measurements were recorded every 20 minutes during the daytime (0700 to 2200 hours) and every 30 minutes during the nighttime hours (2200 to 0700), as preprogrammed into the device. For statistical analyses, diurnal hours were defined as 0800 to 2100 and nocturnal hours were defined as 0000 to 0600. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable mean arterial pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 247 | 251 | 249
millimeters of mercury (mmHg)
  Mean Daytime MAP, Week 16 | -1.30 (0.48) | -0.42 (0.46) | -0.33 (0.47)
  Mean Daytime MAP, Week 26 | -0.51 (0.49) | -0.42 (0.47) | 0.05 (0.48)
  Mean Nighttime MAP, Week 16 | -0.80 (0.56) | -0.59 (0.53) | -1.11 (0.54)
  Mean Nighttime MAP, Week 26 | -0.96 (0.57) | -0.76 (0.54) | -0.50 (0.56)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis — Treatment comparison of mean daytime mean arterial pressure (MAP) at 16 weeks; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-2.22 to 0.28]
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.883, Mixed Models Analysis — Treatment comparison of mean daytime mean arterial pressure (MAP) at 16 weeks; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.32 to 1.13]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.390, Mixed Models Analysis — Treatment comparison of mean daytime mean arterial pressure (MAP) at 26 weeks; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.84 to 0.72]
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.463, Mixed Models Analysis — Treatment comparison of mean daytime mean arterial pressure (MAP) at 26 weeks; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.72 to 0.79]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.671, Mixed Models Analysis — Treatment comparison of mean nighttime mean arterial pressure (MAP) at 16 weeks; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-1.13 to 1.76]
Statistical Analysis 6: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.471, Mixed Models Analysis — Treatment comparison of mean nighttime mean arterial pressure (MAP) at 16 weeks; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.90 to 1.95]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.543, Mixed Models Analysis — Treatment comparison of mean nighttime mean arterial pressure (MAP) at 26 weeks; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.95 to 1.03]
Statistical Analysis 8: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.728, Mixed Models Analysis — Treatment comparison of mean nighttime mean arterial pressure (MAP) at 26 weeks; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.72 to 1.20]

12. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Glycosylated Hemoglobin (HbA1c)
Description: Glycosylated hemoglobin (HbA1c) is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable glycosylated hemoglobin (HbA1c) data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
percentage of HbA1c
  Week 16 | -1.18 (0.06) | -1.04 (0.05) | -0.06 (0.05)
  Week 26 | -1.01 (0.07) | -0.89 (0.06) | -0.02 (0.06)

13. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Fasting Blood Glucose (FBG)
Description: Fasting blood glucose (FBG) is a test to determine how much glucose (sugar) is in a blood sample after an overnight fast. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable fasting blood glucose data.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 249 | 247 | 249
millimoles per liter (mmol/L)
  Week 16 | -2.05 (0.13) | -1.94 (0.13) | -0.30 (0.13)
  Week 26 | -1.67 (0.15) | -1.66 (0.15) | 0.00 (0.15)

14. Secondary Outcome: Percentage of Participants Achieving an Glycosylated Hemoglobin (HbA1c) of <7% or ≤6.5%
Description: Percentages of participants who achieved glycosylated hemoglobin (HbA1c) levels of <7% or ≤6.5% were analyzed with Chi-squared test/Fisher's exact test.
Time Frame: Baseline and 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable glycosylated hemoglobin (HbA1c) data.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
percentage of participants
  HbA1c levels <7.0%, Baseline | 6.8 | 6.7 | 8.0
  HbA1c levels ≤6.5%, Baseline | 0.0 | 0.4 | 0.4
  HbA1c levels <7.0%, Week 16 (n=216, n=234, n=225) | 66.7 | 59.0 | 12.9
  HbA1c levels ≤6.5%, Week 16 (n=216, n=234, n=225) | 45.8 | 36.8 | 6.2
  HbA1c levels <7.0%, Week 26 (n=206, n=226, n=210) | 62.1 | 54.9 | 14.3
  HbA1c levels ≤6.5%, Week 26 (n=206, n=226, n=210) | 38.8 | 35.8 | 5.2

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events at 26 Weeks
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with one or more TEAE is summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo.
Measure: Number; unit: participants
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
participants | 160 | 156 | 162

16. Secondary Outcome: Change From Baseline to 16 and 26 Weeks on Pancreatic Enzymes
Description: Amylase (total and pancreas-derived) and lipase concentrations were measured.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable pancreatic enzyme data.
Measure: Median (Inter-Quartile Range); unit: units per liter
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 214 | 227 | 224
units per liter
  Amylase, Total, Week 16 (n=214, 227, 224) | 6.00 [-2.00 to 13.00] | 5.00 [-3.00 to 14.00] | 0.00 [-6.00 to 7.00]
  Amylase, Total, Week 26 (n=205, 220, 209) | 7.00 [-2.00 to 16.00] | 4.00 [-2.00 to 15.50] | 0.00 [-5.00 to 6.00]
  Amylase, Pancreas-derived, Wk 16 (n=213, 227, 224) | 4.00 [0.00 to 9.00] | 3.00 [-1.00 to 9.00] | 1.00 [-3.50 to 4.00]
  Amylase, Pancreas-derived, Wk 26 (n=204, 220, 209) | 5.00 [1.00 to 10.00] | 3.50 [0.00 to 9.50] | 1.00 [-3.00 to 4.00]
  Lipase, Week 16 (n=214, 227, 224) | 4.00 [-2.00 to 14.00] | 3.00 [-4.00 to 12.00] | -1.00 [-7.00 to 6.00]
  Lipase, Week 26 (n=205, 220, 209) | 6.00 [-1.00 to 14.00] | 5.00 [-3.00 to 13.00] | 0.00 [-6.00 to 5.00]

17. Secondary Outcome: Change From Baseline to 16 and 26 Weeks on Serum Calcitonin
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable serum calcitonin data.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 213 | 223 | 223
picograms per milliliter (pg/mL)
  Week 16 (n=213, n=223, n=223) | -0.30 (1.87) | -0.03 (1.81) | -0.39 (1.24)
  Week 26 (n=202, n=220, n=209) | -0.19 (1.73) | 0.02 (2.04) | -0.05 (2.38)

18. Secondary Outcome: Change From Baseline to 16 Weeks in High-Sensitivity C-Reactive Protein (Hs-CRP)
Time Frame: Baseline, 16 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable High-Sensitivity C-Reactive Protein (hs-CRP) data.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 214 | 228 | 224
milligram per liter (mg/L) | -0.79 (4.91) [-1.27 to 0.14] | -0.20 (7.96) [-1.05 to 0.75] | 0.29 (6.73) [-1.13 to 0.02]

19. Secondary Outcome: Change From Baseline to 16 and 26 Weeks on Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable Fridericia-corrected QT (QTcF) or PR interval change from baseline data.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 248 | 250 | 246
milliseconds (msec)
  QTcF Interval, Week 16 (n=248, n=250, n=246) | -2.31 (0.97) | -0.96 (0.91) | 1.06 (0.93)
  QTcF Interval, Week 26 (n=248, n=250, n=246) | -1.73 (0.96) | -0.93 (0.92) | 1.26 (0.94)
  PR Interval, Week 16 (n=248, n=250, n=244) | 4.96 (0.98) | 3.67 (0.92) | 0.01 (0.95)
  PR Interval, Week 26 (n=248, n=250, n=244) | 3.32 (0.86) | 3.17 (0.81) | -1.98 (0.84)

20. Secondary Outcome: Number of Events of Adjudicated Pancreatitis up to 26 Weeks
Description: The number of adjudicated (by an independent Clinical Endpoint Committee [CEC]) pancreatic events is summarized at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo.
Measure: Number; unit: events
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
events | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events up to 26 Weeks
Description: Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular AEs to be adjudicated include myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo.
Measure: Number; unit: participants
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
participants
  Any cardiovascular event | 1 | 1 | 4
  Any fatal cardiovascular event | 0 | 0 | 0
  Any non-fatal cardiovascular event | 1 | 1 | 4

22. Secondary Outcome: Anti-LY2189265 Antibodies
Description: LY2189265 anti-drug antibodies (ADA) were assessed at baseline, 16 and 26 weeks, and at the safety follow-up visit 4 weeks after study drug discontinuation (30 weeks). The number of participants with initial postbaseline detection of treatment-emergent (defined as a 4-fold increase in the ADA titer from baseline) anti-drug (LY2189265) ADA at each time point were summarized.
Time Frame: Baseline, 16, 26, and 30 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable anti-drug (LY2189265) antibodies (ADA) data.
Measure: Number; unit: participants
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
participants
  Week 16 | 2 | 0 | 0
  Week 26 | 1 | 3 | 0
  Week 30 | 0 | 1 | 0

23. Secondary Outcome: Rate of Hypoglycemic Episodes
Description: Hypoglycemic events (HE) were classified as severe (defined as an HE requiring assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as an HE with typical symptoms of hypoglycemia and a blood glucose level of ≤3.9 millimoles per liter [mmol/L]), asymptomatic (defined as an HE without typical symptoms of hypoglycemia but with a measured blood glucose of ≤3.9 mmol/L), nocturnal (defined as any HE occurring between bedtime and waking with a measured blood glucose of ≤3.9 mmol/L), or non-nocturnal. Hypoglycemia rate per 30 days was summarized at each visit by treatment group. The rate of hypoglycemia was analyzed using a generalized estimation equations model with a negative binomial distribution and a Logit link. Negative binomial mean was adjusted by treatment, visit, and visit by treatment interaction. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo.
Measure: Mean (Standard Deviation); unit: events per participant per 30 days
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
events per participant per 30 days
  Severe | 0 (0) | 0 (0) | 0 (0)
  Documented Symptomatic | 0.14 (0.43) | 0.16 (0.59) | 0.08 (0.39)
  Asymptomatic | 0.17 (0.89) | 0.15 (0.59) | 0.06 (0.25)
  Nocturnal | 0.06 (0.30) | 0.12 (0.64) | 0.03 (0.22)
  Non-nocturnal | 0.29 (0.97) | 0.26 (0.70) | 0.15 (0.44)

24. Secondary Outcome: Change From Baseline to 16 and 26 Weeks in Body Weight
Description: Least Squares (LS) means was calculated using mixed model repeated measures (MMRM) adjusting for baseline, pooled sites, treatment, visit, treatment-by-visit interaction, and the stratified variable of diagnosis of hypertension.
Time Frame: Baseline, 16 and 26 weeks
Population: Participants who received at least one dose of LY2189265 or Placebo with evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Number analyzed (Participants) | 251 | 254 | 250
kilogram (kg)
  Week 16 | -1.84 (0.18) | -0.83 (0.18) | -0.13 (0.18)
  Week 26 | -1.85 (0.23) | -0.86 (0.22) | -0.08 (0.22)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 16 weeks
Statistical Analysis 2: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — Treatment comparison at 16 weeks
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at 26 weeks
Statistical Analysis 4: Comparison: 0.75 Milligram (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — Treatment comparison at 26 weeks

25. Secondary Outcome: Measurement of LY2189265 Drug Concentration for Pharmacokinetics - Area Under the Concentration Time Curve (AUC)
Description: The population mean estimates and standard deviations were calculated for pharmacokinetic parameters (area under the concentration time curve [AUC] at steady state from time zero to 168 hours after study drug administration). Evaluable pharmacokinetic concentrations from the 4, 8, 12, 16, and 26 weeks timepoints were combined and utilized in a population approach to determine the population mean estimate and standard deviation at steady-state.
Time Frame: 4, 8, 12, 16, and 26 weeks
Population: Participants who received at least one dose of LY2189265 with evaluable LY2189265 concentration data.
Measure: Mean (Standard Deviation); unit: nanograms*hour per liter (ng*h/L)
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265
Number analyzed (Participants) | 227 | 235
nanograms*hour per liter (ng*h/L) | 11208 (3744) | 5998 (2003)

ADVERSE EVENTS:
Arm/Group | 1.5 Milligram (mg) LY2189265 | 0.75 Milligram (mg) LY2189265 | Placebo
Serious Adverse Events (participants affected / at risk) | 12/251 | 8/254 | 8/250
Other Adverse Events (participants affected / at risk) | 164/251 | 161/254 | 163/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 Milligram (mg) LY2189265 (N=251) | 0.75 Milligram (mg) LY2189265 (N=254) | Placebo (N=250)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tonic clonic movements (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/121 (1) | 0/123 (0) | 0/119 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/130 (0) | 0/131 (0) | 1/131 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 0/121 (0) | 0/123 (0) | 1/119 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 Milligram (mg) LY2189265 (N=251) | 0.75 Milligram (mg) LY2189265 (N=254) | Placebo (N=250)
Abdominal pain upper (Gastrointestinal disorders) | 11 (13) | 6 (11) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (9) | 12 (12) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 31 (49) | 24 (29) | 20 (29)
Dyspepsia (Gastrointestinal disorders) | 11 (21) | 15 (20) | 6 (8)
Nausea (Gastrointestinal disorders) | 35 (52) | 18 (22) | 16 (24)
Vomiting (Gastrointestinal disorders) | 19 (35) | 11 (12) | 11 (14)
Nasopharyngitis (Infections and infestations) | 23 (23) | 19 (21) | 24 (28)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 8 (12) | 12 (13)
Decreased appetite (Metabolism and nutrition disorders) | 17 (20) | 9 (9) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 12 (14) | 13 (16)
Dizziness (Nervous system disorders) | 13 (20) | 10 (16) | 7 (10)
Headache (Nervous system disorders) | 25 (41) | 21 (28) | 25 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days